CLINICAL TRIAL: NCT04032925
Title: Understanding the Effects of Pressure-controlled Intermittent Coronary Sinus Occlusion Assisted Percutaneous Coronary Intervention on Coronary Physiology and Left Ventricular Performance
Brief Title: The Pressure-controlled Intermittent Coronary Sinus Occlusion on VentrIcular PERformance Study
Acronym: PICSO-ViPER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment trend (COVID-10 pandemic related) - impossible to reach aim target within anticipated timeframe
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Miracor Medical SA (Industry)
Responsible Party: Principal Investigator, Giovanni Luigi De Maria, Primary Investigator, Oxford University Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14338
Record Dates: First submitted 2019-06-03; First posted 2019-07-25 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PICSO therapy Group (Experimental): This will be the only treatment of the PICSO VIPER study. Within this group patients will be randomised to have cycles of 2 minutes of balloon-induced myocardial schema with PICSO device in "ON" vs "OFF" modality.
  Interventions: Device: PICSO

INTERVENTIONS:
Device: PICSO — PICSO therapy is delivered through the PICSO Impulse System, which consists of the PICSO Impulse console and PICSO impulse catheter. The PICSO therapy is delivered in each patient for a minimum of 20 minutes to a maximum of 45 minutes.
  The PICSO Impulse catheter is automatically activated by the PICSO Impulse console. It is inserted in the coronary sinus via femoral vein access. The PICSO Impulse Console cyclically inflates and deflates the balloon at the tip of the PICSO Impulse catheter, generating transient increase in coronary sinus pressure.

SUMMARY:
The PICSO ViPER study is a prospective single centre cohort study of the use of PICSO in patients presenting acute myocardial infarction and impaired function of the left ventricle and candidate to angioplasty the left anterior descending (LAD) coronary artery.

The percutaneous coronary intervention (PCI) procedure will be undertaken in a standard fashion, in accordance with the Oxford University Hospitals NHS Trust (OUHT) departmental guidelines for PCI, and includes the use of pressure wire measurements before and after stent deployment. PICSO treatment will be added on top of the conventional treatment.

The protocol will constitute of 5 main stages (that will all be performed during index angioplasty procedure). The protocol is complete at the end of the angioplasty procedure, and the patient will exit the study at this point. The five stages of the protocol are described below (for details see "Detailed Description"):

* Baseline
* PICSO treatment during pre-dilation
* Stenting with PICSO support
* Post-stent Physiology
* PICSO treatment during post-dilation

DETAILED DESCRIPTION:
In detail, the five stages of the PICSO VIPER study include:

Stage 1: Baseline

* Diagnostic angiography will be performed in the standard manner using appropriate catheters.
* Pre-stenting coronary physiology parameters, namely fractional flow reserve (FFR), coronary flow reserve (CFR) and index of microcirculatory resistance (IMR) will be measured, using a pressure wire, as used for routine clinical measurements in patients undergoing PCI.
* Via a separate arterial access, a conductance catheter will be inserted retrogradely in the left ventricle for baseline measurements of cardiac pump function .
* Baseline blood samples will be withdrawn from the CS (via PICSO balloon) and ascending aorta (via coronary guiding catheter used for revascularization)

Stage 2: PICSO treatment during pre-dilation

* The PICSO device will be deployed as already previously described in the literature.
* Pre-dilation will be performed using an angioplasty balloon at a size determined by the operator, as per standard clinical practice. Balloon will be maintained inflated for a minimum of 1 minute to a maximum of 2 minutes if well tolerated by the patient.
* Balloon inflation will be performed once with the PICSO device activated and once with PICSO device in standby. The order of this will be determined by randomisation via Sequentially Numbered Opaque Sealed Envelopes.
* During each balloon inflation measurements of coronary and cardiac function will be performed and blood samples will be collected exactly as in stage 1.

Stage 3: Stenting with PICSO support

• Stenting is performed as usual clinical practice while the PICSO device is active. The overall duration of PICSO will be no less than 20 minutes, up to a maximum of 45 minutes.

Stage 4: Post-stent Physiology

* Post-stenting coronary and cardiac physiology parameters will be measured using a pressure wire and conductance catheter, respectively.
* Blood samples will be drawn from the CS and the coronary guide catheter as described in stage 1.

Stage 5

* Stent post-dilation will be performed using an angioplasty balloon at a size determined by the operator, as per standard clinical practice. Balloon will be maintained inflated for a minimum of 1 minute to a maximum of 2 minutes if well tolerated by the patient.
* Balloon inflation will be performed in all patients once with the PICSO device activated and once with the PICSO device in standby. The order of this will be the same as in Stage 2 (as determined by Sequentially Numbered Opaque Sealed Envelopes)
* During each balloon inflation measurements will be made of coronary and cardiac physiology parameters and blood samples will be drawn from the CS and the coronary guide catheter as described in stage 1.
* Following this, the participant completes and exits the study.

ELIGIBILITY:
Inclusion Criteria:

* Admission with NSTEMI and considered for coronary angiogram for a view for PCI
* Echocardiographic evidence of at least mild left ventricular systolic impairment (Ejection Fraction < 50%) or regional wall motion abnormalities in LAD territory
* Angiographically proven stenosis of the LAD treated with PCI

Exclusion Criteria:

* Patient referred for surgical revascularization or considered for medical management of coronary disease
* Planned revascularization by mean of balloon angioplasty without stenting
* Patients in whom safety or clinical concerns preclude participation. These would include:

  * Significant left main stem disease
  * Cardiogenic shock and/or haemodynamic instability at the time of enrolment/screening
* Recent PCI or admission with acute coronary syndrome in the previous 3 months before screening/enrolment
* Known anaemia (Hb < 90 g/L)
* Pregnant or breast-feeding females
* History of stroke, TIA or reversible ischaemic neurological disease within last 6 months
* Known severe renal failure (eGFR < 30 ml/min/1.73m2) or history of dialysis or renal transplant
* Previous coronary bypass artery grafting
* Previous PCI to LAD
* Known severe valvular abnormalities
* Use of warfarin
* Presence of pacemaker electrode or medical device in the coronary sinus
* History of inability or, in the opinion of the investigator, anticipated inability to tolerate pharmacologic stress testing (e.g. second- or third-degree AV block without a cardiac pacemaker, severe asthma, resting systolic blood pressure <90mmHg, unstable coronary disease, use of medications which may interfere with the test).
* Unwilling, or unable, to give informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
End-systolic pressure volume relationship (ESPVR) | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Parameter of ventricular physiology and performance
End diastolic pressure volume relationship (EDPVR) | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Parameter of ventricular physiology and performance
Minimum dp/dt | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Parameter of ventricular physiology and performance
Maximum dp/dt | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Parameter of ventricular physiology and performance
Tau | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Parameter of ventricular physiology and performance
Stroke work | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Parameter of ventricular physiology and performance
Pressure-Volume Area (PVA) | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Parameter of ventricular physiology and performance
Cardiac Efficiency | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Parameter of ventricular physiology and performance

SECONDARY OUTCOMES:
Transcoronary gradient of lactates levels | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Cardiac metabolism and energetics
Transcoronary oxygen content | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Cardiac metabolism and energetics
Transcoronary microRNA gradient | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Cardiac metabolism and energetics

OTHER OUTCOMES:
Measurement of IMR | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Coronary microvascular function
Measurement of CFR | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Coronary microvascular function
Measurement of Coronary wedge pressure during balloon occlusion. | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Coronary microvascular function
Time for PICSO deployment | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Safety Endpoint rate of coronary sinus complications: perforation, dissection, thrombosis; time for PICSO deployment / screening time and radiation dose
Screening time for PICSO deployment | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Safety Endpoint rate of coronary sinus complications: perforation, dissection, thrombosis; time for PICSO deployment / screening time and radiation dose
Radiation dose for PICSO deployment | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Safety Endpoint
Rate of coronary sinus perforation | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Safety Endpoint
Rate of coronary sinus dissection | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Safety Endpoint
Rate of coronary sinus thrombosis | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Safety Endpoint
Rate of PICSO failure deployment | At completion of index percutaneous coronary intervention (on average 90 minutes post enrolment)
  Safety Endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Luigi De Maria, MD, PhD, Study Chair — Oxford University Hospitals - NHS Foudation Trust
Locations (1):
- Oxford Heart Centre, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Kirtane AJ, Moses JW. Revascularization in heart failure: the role of percutaneous coronary intervention. Heart Fail Clin. 2007 Apr;3(2):229-35. doi: 10.1016/j.hfc.2007.05.003. PMID 17643923
- [Background] Martinez GJ, Yong AS, Fearon WF, Ng MK. The index of microcirculatory resistance in the physiologic assessment of the coronary microcirculation. Coron Artery Dis. 2015 Aug;26 Suppl 1:e15-26. doi: 10.1097/MCA.0000000000000213. PMID 26247265
- [Background] Lazar HL, Rajaii A, Roberts AJ. Reversal of reperfusion injury after ischemic arrest with pressure-controlled intermittent coronary sinus occlusion. J Thorac Cardiovasc Surg. 1988 Apr;95(4):637-42. PMID 3352298
- [Background] Spaan JA. Mechanical determinants of myocardial perfusion. Basic Res Cardiol. 1995 Mar-Apr;90(2):89-102. doi: 10.1007/BF00789439. No abstract available. PMID 7646422
- [Background] Duncker DJ, Bache RJ. Regulation of coronary blood flow during exercise. Physiol Rev. 2008 Jul;88(3):1009-86. doi: 10.1152/physrev.00045.2006. PMID 18626066
- [Background] Lazar HL. Advantages of pressure-controlled intermittent coronary sinus occlusion over left ventricle-powered coronary sinus retroperfusion. Ann Thorac Surg. 2001 Jan;71(1):402. doi: 10.1016/s0003-4975(00)02036-1. No abstract available. PMID 11216805
- [Background] Martin JS, Byrne JG, Ghez OY, Sayeed-Shah U, Grachev SD, Laurence RG, Cohn LH. LV-powered coronary sinus retroperfusion reduces infarct size in acutely ischemic pigs. Ann Thorac Surg. 2000 Jan;69(1):84-9. doi: 10.1016/s0003-4975(99)00865-6. PMID 10654492
- [Background] Ido A, Hasebe N, Matsuhashi H, Kikuchi K. Coronary sinus occlusion enhances coronary collateral flow and reduces subendocardial ischemia. Am J Physiol Heart Circ Physiol. 2001 Mar;280(3):H1361-7. doi: 10.1152/ajpheart.2001.280.3.H1361. PMID 11179085
- [Background] Mohl W, Mina S, Milasinovic D, Kasahara H, Wei S, Maurer G. Is activation of coronary venous cells the key to cardiac regeneration? Nat Clin Pract Cardiovasc Med. 2008 Sep;5(9):528-30. doi: 10.1038/ncpcardio1298. No abstract available. PMID 18679384
- [Background] Van de Hoef TP, Nolte F, Delewi R, Henriques JP, Spaan JA, Tijssen JG, Siebes M, Wykrzykowska JJ, Stone GW, Piek JJ. Intracoronary hemodynamic effects of pressure-controlled intermittent coronary sinus occlusion (PICSO): results from the First-In-Man Prepare PICSO Study. J Interv Cardiol. 2012 Dec;25(6):549-56. doi: 10.1111/j.1540-8183.2012.00768.x. Epub 2012 Sep 20. PMID 22994798
- [Background] van de Hoef TP, Nijveldt R, van der Ent M, Neunteufl T, Meuwissen M, Khattab A, Berger R, Kuijt WJ, Wykrzykowska J, Tijssen JG, van Rossum AC, Stone GW, Piek JJ. Pressure-controlled intermittent coronary sinus occlusion (PICSO) in acute ST-segment elevation myocardial infarction: results of the Prepare RAMSES safety and feasibility study. EuroIntervention. 2015 May;11(1):37-44. doi: 10.4244/EIJY15M03_10. PMID 25868741
- [Background] De Maria GL, Alkhalil M, Borlotti A, Wolfrum M, Gaughran L, Dall'Armellina E, Langrish JP, Lucking AJ, Choudhury RP, Kharbanda RK, Channon KM, Banning AP. Index of microcirculatory resistance-guided therapy with pressure-controlled intermittent coronary sinus occlusion improves coronary microvascular function and reduces infarct size in patients with ST-elevation myocardial infarction: the Oxford Acute Myocardial Infarction - Pressure-controlled Intermittent Coronary Sinus Occlusion study (OxAMI-PICSO study). EuroIntervention. 2018 Jun 8;14(3):e352-e359. doi: 10.4244/EIJ-D-18-00378. PMID 29792403